CLINICAL TRIAL: NCT05802745
Title: Airway Occlusion Pressure (P0.1) to Predict Extubation Failure in Critically Ill Patients: A Prospective Cohort Study
Brief Title: P0.1 and Extubation Failure in Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cleveland Clinic Abu Dhabi (Other)
Responsible Party: Principal Investigator, Jihad Mallat, Staff Physician, Cleveland Clinic Abu Dhabi
Other Study IDs: A-2023-014
Record Dates: First submitted 2023-03-25; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Weaning Failure; Mechanical Ventilation; Critically Ill
Keywords: Airway occlusion pressure; Extubation failure; Critically Ill patients; Weaning; Mechanical ventilation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Extubation failure: Patients who will require to be re-intubated within 72 hours after extubation.
  Interventions: Other: Reintubation
- Extubation success: Patients who will not require reintubation within 72 hours of extubation.

INTERVENTIONS:
Other: Reintubation — Patients requiring re-intubation for acute respiratory failure.
  Groups: Extubation failure

SUMMARY:
Weaning and extubation are essential steps for the management of critically ill patients when mechanical ventilation (MV) is no longer required. Extubation failure (EF) occurs in approximately 10-30% (1,2) of all patients meeting the readiness criteria and have tolerated a spontaneous breathing trial (SBT). EF is associated with prolonged MV, as well as increased morbidity and mortality (2). Therefore, the early identification of critically ill patients who are likely to experience EF is vital for improved outcomes.

EF can result from different factors (respiratory, metabolic, neuromuscular), particularly cardiac factor, and can be caused by the inability of the respiratory muscle pump to tolerate increases in the cardiac and respiratory load (1,3).

Respiratory drive represents the intensity of the neural stimulus to breathe. In mechanically ventilated patients, it can be abnormally low (i.e., suppressed or insufficient) or abnormally high (i.e., excessive), and thus result in excessively low or high inspiratory effort, leading to potential injury to the respiratory muscles (i.e., myotrauma) (4,5) or to the lungs. A high incidence of abnormal drive (low or high) may explain the high incidence of diaphragm dysfunction at time of separation from mechanical ventilation (6).

Airway occlusion pressure (P0.1) is the drop in airway pressure (Paw) 100 milliseconds after the onset of inspiration during an end-expiratory occlusion of the airway (7). P0.1 measurement is not perceived by the patient and does not influence respiratory pattern. It is, in theory, a reliable measure of respiratory drive because the brevity of the occlusion explains that it is not affected by patient's response to the occlusion and it is independent of respiratory mechanics (8). P0.1 has also been correlated with inspiratory effort (9, 10) and it has been shown that in patients under assisted mechanical ventilation P0.1 might be able to detect potentially excessive inspiratory effort (11).

P0.1 is a non-invasive measure and clinically available at bedside since currently nearly all modern ventilators provide a means of measuring it. Originally, a high P0.1 during a spontaneous breathing trial was associated with failure, suggesting that a high respiratory drive could predict weaning failure. However, only a few and old clinical studies investigated the association between P0.1 and extubation failure (EF) and were not conclusive (12,13). We hypothesized that patients with EF would have increased P0.1 values during spontaneous breathing trial (SBT). Therefore, the aims of our study will be to (1) to evaluate the ability of changes in P0.1 (Delta-P0.1) during SBT to predict EF and (2) to assess if Delta-P0.1 is an independent predictor of EF.

DETAILED DESCRIPTION:
Weaning protocol SBTs will be performed in semirecumbent patients on Pressure Support Ventilation (PSV) mode with inspiratory pressure of 5 cmH2O and positive-end-expiratory pressure (PEEP) of 5 cmH2O as per ICU protocol. Inspiratory oxygen fraction (FiO2) will be adjusted for the achievement of an arterial oxygen saturation value > 90%, as measured by pulse oximetry. The SBT duration will be 30 minutes as per ICU protocol. The criteria that will be used for poor SBT tolerance are: (1) diaphoresis; (2) use of accessory respiratory muscles; (3) RR > 35/min; (4) oxygen saturation by pulse oximetry < 90% with FiO2 ≥ 50%; (5) HR > 140/min or greater than a 20% increase from baseline; (6) Systolic blood pressure >180 mmHg or <90 mmHg; (7) development of cardiac arrhythmias; and/or low level of consciousness.

The decision to stop SBT will be made by the physicians. Patients who will fail SBT will be shifted to their previous ventilator mode and not be enrolled in the study.

Patients who will complete the SBT will be extubated and followed-up for 72 hours. The medical team (physician, nurse, and respiratory therapist) involved in the extubation decision will be blinded to the P0.1 results. EF will be diagnosed if the patient is extubated but required reintubation within the following 72 hours. Criteria for acute respiratory failure after extubation are the development of at least one of the following: (a) respiratory acidosis with pH < 7.32 and arterial CO2 pressure (PaCO2) > 45 mmHg; (b) arterial oxygen saturation < 90% with FiO2 > 0.5; (c) RR > 35/min; (d) clinical signs of respiratory fatigue.

The management of post-extubation respiratory failure will not be protocolized and will be left to the physician's discretion.

Ventilatory, including P0.1 and hemodynamic parameters, including EtCO2 will be recorded as the average of at least three measurements immediately before SBT, during SBT, and at 30 minutes after SBT initiation. Arterial and central venous blood gas (if central line present) will be measured immediately before SBT and at 30 minutes after SBT initiation.

ELIGIBILITY:
Inclusion Criteria:

- All patients aged 18 years or older who received mechanical ventilation for at least 48 hours and satisfied the weaning criteria will be eligible for enrollment.

The readiness-to-wean criteria that will be employed are: (1) the resolution or improvement of the underlying cause of respiratory failure for which the patient was intubated; (2) hemodynamic stability, defined as heart rate (HR) < 140/min and systolic blood pressure between 90 and 160 mmHg with no or minimal doses of vasopressors; (3) stable respiratory status, defined as oxygen saturation > 90% with fraction of inspired oxygen (FiO2) ≤ 0.5 and positive end expiratory-pressure (PEEP) ≤8 cmH2O, respiratory rate (RR) ≤ 35/min, spontaneous tidal volume (Vt) > 5 mL/kg, and no significant respiratory acidosis; (4) adequate mental status, and (5) adequate cough.

Exclusion Criteria:

* Presence of tracheostomy
* Do-not-reintubate orders
* pregnancy
* Absence of informed consent
* Spontaneous breathing trial failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with invasive mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Extubation failure | Within 72 hours after extubation.
  to evaluate the ability of changes in P01 (Delta-P0.1) during SBT to predict extubation failure after 72 hours of extubation.

SECONDARY OUTCOMES:
Delta-P01 as independent factor of extubation failure | Within 72 hours after extubation.
  To assess if Delta- P0.1 during SBT is an independent predictor of extubation failure
Extubation failure | 7 days after extubation
  Association between Delta-P0.1 and extubation failure after 7 days of extubation

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Mallat, MD, PhD, Principal Investigator — Cleveland Clinic Abu Dhabi
Locations (3):
- France (3):
  - Amiens University Hospital, Amiens
  - Centre Hospitalier d'Arras, Arras
  - Dijon University Hospital, Dijon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Result] Thille AW, Richard JC, Brochard L. The decision to extubate in the intensive care unit. Am J Respir Crit Care Med. 2013 Jun 15;187(12):1294-302. doi: 10.1164/rccm.201208-1523CI. PMID 23641924
- [Result] MacIntyre N. Discontinuing mechanical ventilatory support. Chest. 2007 Sep;132(3):1049-56. doi: 10.1378/chest.06-2862. PMID 17873200
- [Result] Goligher EC, Dres M, Fan E, Rubenfeld GD, Scales DC, Herridge MS, Vorona S, Sklar MC, Rittayamai N, Lanys A, Murray A, Brace D, Urrea C, Reid WD, Tomlinson G, Slutsky AS, Kavanagh BP, Brochard LJ, Ferguson ND. Mechanical Ventilation-induced Diaphragm Atrophy Strongly Impacts Clinical Outcomes. Am J Respir Crit Care Med. 2018 Jan 15;197(2):204-213. doi: 10.1164/rccm.201703-0536OC. PMID 28930478
- [Result] Goligher EC, Brochard LJ, Reid WD, Fan E, Saarela O, Slutsky AS, Kavanagh BP, Rubenfeld GD, Ferguson ND. Diaphragmatic myotrauma: a mediator of prolonged ventilation and poor patient outcomes in acute respiratory failure. Lancet Respir Med. 2019 Jan;7(1):90-98. doi: 10.1016/S2213-2600(18)30366-7. Epub 2018 Nov 16. PMID 30455078
- [Result] Dres M, Dube BP, Mayaux J, Delemazure J, Reuter D, Brochard L, Similowski T, Demoule A. Coexistence and Impact of Limb Muscle and Diaphragm Weakness at Time of Liberation from Mechanical Ventilation in Medical Intensive Care Unit Patients. Am J Respir Crit Care Med. 2017 Jan 1;195(1):57-66. doi: 10.1164/rccm.201602-0367OC. PMID 27310484
- [Result] Telias I, Damiani F, Brochard L. The airway occlusion pressure (P0.1) to monitor respiratory drive during mechanical ventilation: increasing awareness of a not-so-new problem. Intensive Care Med. 2018 Sep;44(9):1532-1535. doi: 10.1007/s00134-018-5045-8. Epub 2018 Jan 19. No abstract available. PMID 29350241
- [Result] Whitelaw WA, Derenne JP, Milic-Emili J. Occlusion pressure as a measure of respiratory center output in conscious man. Respir Physiol. 1975 Mar;23(2):181-99. doi: 10.1016/0034-5687(75)90059-6. PMID 1144940
- [Result] Alberti A, Gallo F, Fongaro A, Valenti S, Rossi A. P0.1 is a useful parameter in setting the level of pressure support ventilation. Intensive Care Med. 1995 Jul;21(7):547-53. doi: 10.1007/BF01700158. PMID 7593895
- [Result] Mancebo J, Albaladejo P, Touchard D, Bak E, Subirana M, Lemaire F, Harf A, Brochard L. Airway occlusion pressure to titrate positive end-expiratory pressure in patients with dynamic hyperinflation. Anesthesiology. 2000 Jul;93(1):81-90. doi: 10.1097/00000542-200007000-00016. PMID 10861149
- [Result] Rittayamai N, Beloncle F, Goligher EC, Chen L, Mancebo J, Richard JM, Brochard L. Effect of inspiratory synchronization during pressure-controlled ventilation on lung distension and inspiratory effort. Ann Intensive Care. 2017 Oct 6;7(1):100. doi: 10.1186/s13613-017-0324-z. PMID 28986852
- [Result] Sassoon CS, Te TT, Mahutte CK, Light RW. Airway occlusion pressure. An important indicator for successful weaning in patients with chronic obstructive pulmonary disease. Am Rev Respir Dis. 1987 Jan;135(1):107-13. doi: 10.1164/arrd.1987.135.1.107. PMID 3800139
- [Result] Fernandez R, Raurich JM, Mut T, Blanco J, Santos A, Villagra A. Extubation failure: diagnostic value of occlusion pressure (P0.1) and P0.1-derived parameters. Intensive Care Med. 2004 Feb;30(2):234-240. doi: 10.1007/s00134-003-2070-y. Epub 2003 Nov 8. PMID 14608459